CLINICAL TRIAL: NCT03551106
Title: Can an E-learning Module Improve Prescriptions of Laboratory Examens by Postgraduate Medical Students?
Brief Title: E-learning Module to Improve Laboratory Prescriptions
Acronym: CLAB1
Status: Completed | Type: Observational
Sponsor: Hôpital du Valais (Other)
Responsible Party: Sponsor
Other Study IDs: CLAB1
Record Dates: First submitted 2018-04-25; First posted 2018-06-11 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Learning
Keywords: e-learning; web based learning module

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Web based learning module: Laboratory prescriptions made by postgraduate students who were enrolled to follow the web based modules
  Interventions: Other: Web based learning module

INTERVENTIONS:
Other: Web based learning module — Web based learning module available on a especially designed website

SUMMARY:
Objective: To evaluate the effectiveness of a web based learning module in the prescription of laboratory examens by postgraduate medical students.

Background: The internal medicine service of Valais encounters several prescription issues such as overprescription of blood iron or transferrin level determination and too rare D vitamine level.

Methods: The investigators will introduce postgraduate medical students to a single use e-learning module about common deficiencies in hospitalized patients. A quick test will be performed before and after the module, then at 2 and 4 months. Efficiency will be determined by the analysis of the median number of prescriptions of blood iron, transferrin and D vitamine levels 6 months before the module then monthly until completion of the study . It is planned to recruit between 40 and 55 students.

Outcome: The investigators will evaluate efficiency of the web based learning module by analysing the prescription rate 5 months before and 5 months after the intervention. Second outcome will be testing of the efficiency over time by monthly analysis of the prescriptions and results at the test.

DETAILED DESCRIPTION:
The internal medicine in Valais (switzerland) service encounters several prescription issues partially caused by semi-automatic informatized software. The more often students are not aware of the costs inherent to unuseful laboratory examens and use the quickest way. Furthermore several older students still use prior recommendations for the determination of patient deficiency status. The investigators wish to determine if a web-based instruction module can improve practice and persist over time.

Objective: To evaluate the effectiveness of a web based learning module in the prescription of laboratory examens by postgraduate medical students.

Methods: A website will be especially designed for the purpose. All postgraduate medical students of the internal medicine service will be introduced to the e-learning module as part of routine medical care. Preceding and following this exposure the investigators will measure how well the students perform to a comprehensive 10-item assessment tool designed by experienced internists in the Department.

40 to 55 students are expected to participate in the study. A quick test will be performed before and after the module, then at 2 and 4 months. Efficiency will be determined by the analysis of the median number of prescriptions of blood iron, transferrin and D vitamine levels 5 months before the module then at the completion of the study.

Pre and post-test will be used to evaluate the efficiency of the short learning module, and test at 2 and 4 months to estimate the persistence of these results over time.

The prescription of B9 and B12 levels as well as the management of the obtained results will also be analysed.

Limitations: This design does not incorporate a comparison group, because of the insufficient number of students for this method. Multicenter study with comparison group will be performed if results are promising.

ELIGIBILITY:
Inclusion Criteria:

* Post graduate student
* Enrolled in our internal medicine service

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All of the postgraduate medical students of the internal medicine service in Valais.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Prescription efficiency | 4 months
  We will evaluate efficiency of the web based learning module by analysing the prescription rate 4 months after the intervention

SECONDARY OUTCOMES:
Mid term impact on prescription | 1 month, 2 months, 3 months and 4 months
  Efficiency over time by monthly analysis of the prescriptions. Prescriptions rate will be evaluated monthly in order to evaluate the persistency of the module.
Web based module validity | 1 day, 2 months and 4 months
  Web based module efficiency over time: using a 10-item assessment tool at day 1 (before and after reading of the module) then 2 months and 4 months after the beginning of the study.
  Obtained score will be on a scale of 0 to 10, each correct answer allowing 1 point

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Auguste PETIGNAT, MD, Study Director — Hôpitaux du Valais; Damien LE PEILLET, MD, Principal Investigator — Hôpitaux du Valais
Locations (1):
- Hopital du Valais, Sion, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Keijsers CJ, van Doorn AB, van Kalles A, de Wildt DJ, Brouwers JR, van de Kamp HJ, Jansen PA. Structured pharmaceutical analysis of the Systematic Tool to Reduce Inappropriate Prescribing is an effective method for final-year medical students to improve polypharmacy skills: a randomized controlled trial. J Am Geriatr Soc. 2014 Jul;62(7):1353-9. doi: 10.1111/jgs.12884. Epub 2014 Jun 10. PMID 24916615
- [Result] Maxwell S, Mucklow J. e-Learning initiatives to support prescribing. Br J Clin Pharmacol. 2012 Oct;74(4):621-31. doi: 10.1111/j.1365-2125.2012.04300.x. PMID 22509885